CLINICAL TRIAL: NCT07122609
Title: A Study of Pirtobrutinib in Combination With Rituximab, Gemcitabine, Oxaliplatin With or Without Polatuzumab Vedotin (Pirto-R-GemOx±Pola) in Covalent BTK Inhibitor-Pretreated Relapsed/Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Brief Title: Pirtobrutinib in Combination With Rituximab, Gemcitabine, Oxaliplatin With or Without Polatuzumab Vedotin in Covalent BTK Inhibitor-Pretreated Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, First Deputy Director of Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: pirto-R-Gemox
Record Dates: First submitted 2025-07-27; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Relapsed and Refractory DLBCL
MeSH Terms: conditions — Recurrence | interventions — pirtobrutinib; polatuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- pirtobrutinib+R-GemOx with or without polatuzumab vedotin (Experimental): DLBCL patients will receive Pirto-R-GemOx for a total of 6 treatment cycles (21days per cycle). Patient who is CD79b positive and has not previously received polatuzumab Vedotin will combine with polatuzumab Vedotin.The efficacy will be evaluated every 3 cycles, young patients with CR will receive ASCT, CR patients who do not undergo ASCT or PR patients will continued for 3 cycles.If the efficacy is evaluated as CR or PR after 6 cycles, then ASCT for young patients, and lenalidomide maintenance treatment for elderly patients for 2 years (25mg, day 1-21, Q4W). ctDNA testing will be performed at baseline、before the second course、and at the end of treatment.
  Interventions: Drug: Pirtobrutinib; Drug: R-GemOx; Drug: Polatuzumab Vedotin

INTERVENTIONS:
Drug: Pirtobrutinib — Dose:200mg，d1-21
  Other Names: LOXO-305
Drug: R-GemOx — Dose: Rituximab: 375mg/m2, d1; Gemcitabine: 1000mg/m2, d2; Oxaliplatin:100mg/m2, d2
Drug: Polatuzumab Vedotin — Dose: 1.8mg/kg，iv，d1 (For patient who is CD79b positive and has not previously received polatuzumab Vedotin)

SUMMARY:
This is a prospective, single arm trial in patients with ≥ 18 years with relapsed and refractory DLBCL. Aim of this study is to evaluate the efficacy and safety of pirtobrutinib in combination with rituximab, gemcitabine, and oxaliplatin with or without polatuzumab vedotin (Pirto-R-GemOx±pola) in patients with relapsed/refractory diffuse large B-cell lymphoma (R/R DLBCL) previously treated with covalent BTK inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed DLBCL (2016 WHO criteria) of MCD, BN2, N1 subtypes, double-expressor, intravascular large B-cell lymphoma, or other BTK-sensitive subtypes
* Disease progression/relapse after covalent BTK inhibitor therapy
* ≥1 measurable lesion (nodal >15mm/extranodal >10mm) on PET/CT within 28 days
* Eastern Cooperative Oncology Group (ECOG) 0-2
* age ≥18 years
* Adequate organ function:

ANC ≥0.5×10⁹/L ；Platelets ≥50×10⁹/L (transfusion-independent)；Bilirubin ≤1.5×ULN; ALT/AST ≤2.5×ULN；Cr ≤1.5×ULN or CrCl ≥30mL/min；LVEF ≥50% (NYHA class <III)

* Life expectancy >3 months
* Sign the written ICF, and be able to comply with the visits and related procedures stipulated in the protocol;
* Female subjects of childbearing potential or male subjects with female partners of childbearing potential must use effective contraception throughout the treatment period and for 90 days after the last treatment.

Exclusion Criteria:

* DLBCL with central nervous system (CNS) or meningeal involvement
* Histologically transformed DLBCL
* Contraindications or hypersensitivity to any drug in the combination regimen
* Major surgery within 4 weeks prior to treatment (excluding vascular access placement or biopsy)
* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's judgment, may compromise patient safety or compliance with study procedures
* Poorly controlled cardiac clinical symptoms or diseases, including:

  i. NYHA Class II or higher heart failure ii. Unstable angina iii. Myocardial infarction within 1 year iv. Clinically significant supraventricular or ventricular arrhythmias requiring treatment/intervention
* Active hemorrhage
* Poorly controlled systemic bacterial, viral, fungal, or parasitic infections (excluding fungal nail infections), or other clinically significant active diseases that render patients unsuitable for trial participation per investigator assessment
* Patients with:Active chronic hepatitis B or C.Positive HBsAg and/or HBcAb or HCV antibodies at screening must demonstrate HBV DNA ≤2,500 copies/mL (or 500 IU/mL) to exclude active HBV/HCV infection requiring treatment.HBsAg/HBcAb-positive patients must receive antiviral prophylaxis.

HIV-infected patients and/or AIDS patients

* Inability to swallow tablets, malabsorption syndrome, or any gastrointestinal disorder/ dysfunction that may impair drug absorption
* Lactating or pregnant women
* Psychiatric disorders or inability to provide informed consent
* Any other condition deemed unsuitable for study participation by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-08-05 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
complete response rate(CRR) | Up to 6 cycles (each cycle is 21 days)
  CRR after treated by pirto-R-GemOx±pola

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to 6 cycles (each cycle is 21 days) ± pola
  ORR after treated by pirto-R-GemOx
Progression-free survival (PFS) | Up to 6 cycles (each cycle is 21 days)
  PFS after treated by pirto-R-GemOx±pola
Overall Survival (OS) | up to 6 cycles(each cycle is 21 days)
  OS after treated by pirto-R-GemOx±pola
undetectable MRD rate | Up to 6 cycles (each cycle is 21 days) ± pola
  undetectable MRD rate after treated by pirto-R-GemOx

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Professor, Principal Investigator — Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine
Locations (1):
- Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No